CLINICAL TRIAL: NCT03985995
Title: Pain Response to Cannabidiol in Induced Acute Nociceptive Pain, Allodynia and Hyperalgesia By Using a Model Mimicking Acute Pain in Healthy Adults
Acronym: CANAB I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019-00839; qu18Ruppen2
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Pain Sensation; Hyperalgesia; Allodynia
Keywords: Cannabidiol (CBD)
MeSH Terms: conditions — Hyperalgesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBD 800 mg p.o. (Active Comparator): The study Investigational Medical Product (IMP) is a cannabidiol solution 100 mg/ml 8 ml in single-dose containers for per os administration.
  Interventions: Drug: CBD 800 mg p.o
- Placebo p.o. (Placebo Comparator): Participants in the control arm will be receiving a single dose of oral placebo solution 8 ml matched to the active comparator.
  Interventions: Drug: Placebo p.o

INTERVENTIONS:
Drug: CBD 800 mg p.o — cannabidiol solution 100 mg/ml 8 ml in single-dose containers for per os administration. After a washout period of at least two weeks, the treatment group will be receiving a single-dose of the placebo solution 8 ml as a second intervention.
  Arms: CBD 800 mg p.o.
Drug: Placebo p.o — single dose of oral placebo solution 8 ml matched to the IMP. After a washout period of at least two weeks, the control intervention group will be receiving the cannabidiol solution 100 mg/ml 8 ml as a second intervention.
  Arms: Placebo p.o.

SUMMARY:
This study is to investigate the effect of CBD on acute pain in healthy volunteers in a well-established acute pain model.

DETAILED DESCRIPTION:
There are no studies investigating Cannabidiol (CBD) in an acute pain model in human beings. This is however of great clinical value because:

1. Patients are often treated insufficiently with the commonly used analgesics in acute pain therapy or the available selection of analgesics is limited by their contraindications and side-effects.
2. CBD could be an option to optimize pain therapy if the pain relief is not satisfactory.
3. CBD in contrast to ∆9-tetrahydrocannabinol (THC) has only few side effects and due to a possible dose reduction of other analgesics patients might benefit from a better side-effect profile.

This study is to investigate the effect of CBD on acute pain in healthy volunteers in a well-established acute pain model.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* BMI between 18.5 until 25 kg/m2
* Able to understand the study and the NRS scale
* Able to give informed consent

Exclusion Criteria:

* Regular consumption of cannabinoids or other drugs / substances
* Regular intake of medications potentially interfering with pain sensation (analgesics, antihistamines, calcium and potassium channel blockers, serotonin / noradrenaline reuptake inhibitors, corticosteroids)
* Neuropathy
* Chronic pain
* Neuromuscular disease
* Psychiatric disease
* Known or suspected kidney or liver disease
* Pregnancy/ Lactation
* Allergy / hypersensitivity to cannabidiol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Change in pain (numeric rating scale (NRS): 0 = no pain and 10 = maximum tolerable pain) | pain will be assessed every 10 minutes using the NRS from minute 70 to 130
  Change in pain for 60 min (from minute 70 to 130) after inducing defined pain in an experimental setting (Koppert model). 2 microdialysis catheters are inserted into intradermal surface of forearm and attached to a constant current stimulator.

SECONDARY OUTCOMES:
Change in area of hyperalgesia (cm) | from minute 70 to 130
  Change in area of hyperalgesia (from minute 70 to 130) after inducing a defined pain in an experimental setting (Koppert model). Immediately after every pain rating the area of pinprick hyperalgesia is determined using a 256 MilliNewton (mN) von Frey Filament. The von Frey Filament will be moved towards the site of stimulation in 0.5 cm increments until the subject reports increased pain sensations from the von Frey filament (hyperalgesia). To create an area from these linear measurements, the assumption is made, that this field has the shape of an ellipse. The area is calculated using the formula 1/4πD·d.
Change in area of allodynia (cm) | from minute 70 to 130
  Change in area of allodynia (from minute 70 to 130) after inducing a defined pain in an experimental setting (Koppert model). Immediately after every pain rating the area of allodynia is determined using a dry cotton swab. The Cotton swab will be moved towards the site of stimulation in 0.5 cm increments until the subject reports an unpleasant "rougher" sensation from the cotton swab (allodynia). To create an area from these linear measurements, the assumption is made, that this field has the shape of an ellipse. The area is calculated using the formula 1/4πD·d.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Schneider, Dr. med, Principal Investigator — Department of Anaesthesiology, University Hospital of Basel
Locations (1):
- Department of Anaesthesiology, University Hospital of Basel (USB), Basel, Switzerland

REFERENCES:
- [Derived] Schneider T, Zurbriggen L, Dieterle M, Mauermann E, Frei P, Mercer-Chalmers-Bender K, Ruppen W. Pain response to cannabidiol in induced acute nociceptive pain, allodynia, and hyperalgesia by using a model mimicking acute pain in healthy adults in a randomized trial (CANAB I). Pain. 2022 Jan 1;163(1):e62-e71. doi: 10.1097/j.pain.0000000000002310. PMID 34086631